CLINICAL TRIAL: NCT02401659
Title: Importance of Patient´s Satisfaction With Telemedicine Based on Monitoring Systems
Acronym: VALIOSA
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: T431 v 2.0
Record Dates: First submitted 2015-03-17; First posted 2015-03-30 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-11

CONDITIONS: Arrythmia
Keywords: remote monitoring; satisfaction; telemonitoring; quality of life
MeSH Terms: conditions — Arrhythmias, Cardiac; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- naïve with CareLink: patients with a first implant of an implanted cardiac device naïve in CareLink or patients with a refill who have not used CareLink until the implant
  Interventions: Device: CareLinK
- users of CareLink: patients with an implanted cardiac device who have used CareLink for more than one year
  Interventions: Device: CareLinK

INTERVENTIONS:
Device: CareLinK

SUMMARY:
Valiosa is a national, multicenter and prospective post market study. The objectives of the study are to generate and validate an instrument to evaluate patient and clinician's satisfaction with remote monitoring and to create awareness of the importance of remote monitoring among patients, physicians and decision makers.

ELIGIBILITY:
Inclusion Criteria:

1. Patients- naïve in CareLink®:

   * First implant patients, who initiate in CareLink®
   * Replacements patients who initiate in CareLink.
2. Long term users in CareLink®: patients in CareLink for more than a year.
3. Both male and female
4. More than 18 years old.
5. Be at the disposal of using CareLink monitoring system.
6. Complete informed consent and accept the conditions of CareLink system.

Exclusion Criteria:

1. Less than 18 years old
2. Suffer from any menthal pathology who prevents the patient to collaborate in the study.
3. Be unable to understand or answer questionnaires in Spanish.
4. Deny to continue in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an implantable cardiac device and using CareLink® program for the remote monitoring of the device.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2014-05; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Satisfaction with telemedicine measured by the questionnaire in evaluation | 12 months

SECONDARY OUTCOMES:
Satisfaction with medical treatment measured by visual analog scale | 12 months
Quality of Life measured by SF-36 | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Basque Country
  - Hospital Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid